CLINICAL TRIAL: NCT07263659
Title: Virtual Reality Reduces Pre-Procedural Anxiety in TEER Pa-tients, But Timing Seems Crucial
Brief Title: Virtual Reality Reduces Pre-Procedural Anxiety in TEER Patients, But Timing Seems Crucial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abby Geerlings (Other)
Responsible Party: Sponsor-Investigator, Abby Geerlings, PhD/MD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: W21_185#21.239
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Anxiety; Mitral Regurgitation; Tricuspid Regurgitation (TR); Mitraclip; TriClip; Virtual Reality
Keywords: Virtual Reality; Mitraclip; Triclip
MeSH Terms: conditions — Anxiety Disorders; Mitral Valve Insufficiency; Tricuspid Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: articipants will be randomly assigned to one of two parallel groups: a control group receiving standard pre-procedural information and an intervention group receiving standard information supplemented with a virtual reality (VR) educational session. Outcomes will be compared between groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group - Standard Education (No Intervention): Participants in this group will receive standard pre-procedural education according to the hospital's routine practice. This includes verbal and written information provided by the healthcare team about the MitraClip or TricuspidClip procedure, preparation, and aftercare.
- VR Group - Standard Education plus Virtual Reality (VR) (Active Comparator): Participants in this group will receive the same standard pre-procedural education as the control group, supplemented with an immersive virtual reality (VR) experience. The VR session provides a visual and interactive explanation of the procedure and hospital environment to enhance understanding, reduce anxiety, and improve the overall patient experience.
  Interventions: Behavioral: Standard Education plus Virtual Reality (VR)

INTERVENTIONS:
Behavioral: Standard Education plus Virtual Reality (VR) — Participants in this group will receive the same standard pre-procedural education as the control group, supplemented with an immersive virtual reality (VR) experience. The VR session provides a visual and interactive explanation of the procedure and hospital environment to enhance understanding, reduce anxiety, and improve the overall patient experience.
  Other Names: Virtual reality
  Arms: VR Group - Standard Education plus Virtual Reality (VR)

SUMMARY:
This study aims to evaluate the effect of adding virtual reality (VR) education to standard pre-procedural information on anxiety levels in patients scheduled for MitraClip or TricuspidClip procedures. Participants will receive either standard pre-procedural information or standard information supplemented with a VR experience that explains the procedure and hospital environment. The main outcomes will include changes in patient-reported anxiety before and after the procedure. The goal of this study is to determine whether the use of VR can improve patient understanding, reduce procedural anxiety, and enhance overall well-being

ELIGIBILITY:
Inclusion Criteria:

* Adults scheduled for elective mitral (M-TEER) or tricuspid (T-TEER) transcatheter edge-to-edge repair procedures.

Exclusion Criteria:

* Insufficient proficiency in Dutch.
* Severe visual or auditory impairment that would prevent full engagement with the VR content.
* Any mental or physical condition that, in the judgment of the clinical team, significantly interferes with participation (e.g., advanced cognitive decline, acute psychological distress, or inability to tolerate wearing a VR headset).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Pre-procedural anxiety | 1 week prior to procedure
  Change in state anxiety (S-STAI score) immediately after patient education (VR intervention vs. standard verbal education) and onw week prior to the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data will be made available to researchers upon reasonable request after publication of the main results.